CLINICAL TRIAL: NCT06807606
Title: Optimized CBT for Pts With High-risk Hematologic Malignancies Who Have Relapsed After First ASCT
Brief Title: Optimized Cord Blood Transplantation for the Treatment of Patients With High-risk Hematologic Malignancies Who Have Relapsed After First Allogeneic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1605; NCI-2025-00794 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Thiotepa; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimized CBT (Experimental): Participants enrollment on trial will be determined by consultation with the physicians of the SCT Service.
  Interventions: Drug: Drugs Cyclophosphamide; Drug: Fludarabine; Drug: Thiotepa; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Drugs Cyclophosphamide — Given as standard of care treatment through IV infusion
Drug: Fludarabine — Given as standard of care treatment through IV infusion
Drug: Thiotepa — Given as standard of care treatment through IV infusion
Drug: Tacrolimus — Given as standard of care treatment through IV infusion
Drug: Mycophenolate mofetil — Given as standard of care treatment through IV infusion

SUMMARY:
The goal of this clinical research study is to learn if intermediate-intensity conditioning therapy followed by a cord blood transplant can help to control high-risk hematological malignancies in patients who need a second allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate 1-year overall survival (OS) following CBT with intermediate dose intensity conditioning for patients in need of a second allogeneic stem cell transplantation.

Secondary Objectives:

Speed and success of neutrophil and platelet engraftment. Incidences of graft failure.

• Incidence of day 100 grade II-IV and III-IV aGVHD and day 180 grades II-IV and III-IV aGVHD.

Incidence of 1-year, 2-year, and 3-year cGVHD.

Incidence of TRM (100 days, 6 months, 1 and 2 years).

The probabilities of relapse, OS, PFS, and GRFS at 1 year, 2, and 3 years as listed in the secondary endpoints in section 2.2.

Correlative laboratory studies investigating graft versus leukemia biology.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 0-60 y/o at the time of consent. Adult is defined as patients 18 years of age or older at the time of consent.
2. Patient must have relapsed >100 days since first transplant.
3. Diagnosis and Disease Status:

   a. Acute myelogenous leukemia (AML): i. Patients in morphologic remission (<5% blasts) at the time of transplant, with or without persistent cytogenetic, flow cytometric, or molecular aberrations, or those with hypocellular marrows at time of transplant, are eligible. b. Acute lymphoblastic leukemia (ALL): i. Patients in morphologic remission with less than 5% blasts at time of transplant, with or without persistent cytogenetic, flow cytometric or molecular aberrations, or those or who have hypocellular bone marrows, are eligible. c. Other acute leukemias: i. Acute leukemias of ambiguous lineage or mixed phenotype in morphologic remission with less than 5% blasts at time of transplant, with or without persistent cytogenetic, flow cytometric or molecular aberrations, or those who have hypocellular bone marrows, are eligible. d. Myelodysplastic Syndromes (MDS) or CMML without myelofibrosis. i. Includes MDS with any IPSS risk category.
4. Prior treatment:

   a. To be eligible for this study, patients need to have received one prior allogeneic stem cell transplantation.
5. Karnofsky score equal or greater than 70% for patients aged 16 years and older or Lansky score equal or greater than 70% for patients less than 16 years old (See Appendix B; inpatient Leukemia service transfers without discharge are acceptable provided patient has equivalent KPS as if were outpatient).
6. Renal and Liver function:

   1. Calculated creatinine clearance > 50 ml/min.
   2. Bilirubin < 2 mg/dL (unless benign congenital hyperbilirubinemia or hemolysis).
   3. ALT < 5 x upper limit of normal (ULN).
7. Pulmonary function: corrected diffusion capacity of the lung for carbon monoxide (DLCO) > 60% predicted. This criteria is waived for patients who are developmentally unable to complete pulmonary function test.
8. Left ventricular ejection fraction (MOD-bp) > 50%.
9. Graft Criteria:

   1. Two CB units will be selected according to the current MDACC CB unit selection algorithm.
   2. High resolution 8-allele HLA typing and recipient HLA antibody profile will be performed.
   3. Unit selection will occur based on HLA-match, total nucleated cell (TNC), and CD34+ cell dose adjusted per patient body weight.
   4. The bank of origin will also be considered.
   5. Donor-specific HLA antibodies, if present, will also be taken into consideration.
   6. Each CB unit must be at least 3/8 HLA-matched to the patient considering high-resolution 8-allele HLA typing.
   7. Each CB unit will be required to have a cryopreserved TNC dose of at least 1.5 x 107 TNC/ recipient body weight (TNC/ kg).
   8. Each CB unit will be required to have a cryopreserved CD34+ cell dose of at least 1.0 x 105 CD34+ cells/ recipient body weight (CD34+ cells/kg).
   9. A minimum of one unit will be reserved as a backup graft.
   10. Each CB unit will be required to be cryopreserved in standard cryovolume. (24- 27 ml/s per unit) and be red blood cell depleted.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Warren Fingrut, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org